CLINICAL TRIAL: NCT04153604
Title: Doxycycline for the Prevention of Spontaneous Bacterial Peritonitis
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 061.PHA.2019.D
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cirrhosis; Spontaneous Bacterial Peritonitis
MeSH Terms: conditions — Fibrosis | interventions — Doxycycline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: doxycycline — a tetracycline antibiotic that fights bacteria in the body.

SUMMARY:
The utilization of doxycycline for SBP prophylaxis is a novel practice at MDMC. Therefore, an assessment of safety and efficacy is needed in order to generalize this practice. The publication of this study can potentially introduce a new alternative to guideline-directed therapies for secondary prevention of SBP. Doxycycline is non-inferior to guideline-directed therapies regarding safety and efficacy in primary and secondary prophylaxis for SBP.

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is a common and serious complication in cirrhotic patients with a reported mortality rate of 20 to 30%.1-3 A SBP diagnosis requires abdominal paracentesis and is made in the presence of an elevated ascitic fluid absolute polymorphonuclear leukocyte (PMN) count without an evident intra-abdominal, surgically treatable source of infection.2,3 Common pathogens associated with SBP are Gram-negative colonic organisms. However, in recent years, Gram-positive pathogens have become more common, suggesting the need to evaluate SBP management.1,4-6 The recurrence rate of SBP after an initial episode has been reported to be as high as 70%.1-3 Currently, the American Association for the Study of Liver Disease (AASLD) and European Association for the Study of the Liver (EASL) guidelines recommend the use of sulfamethoxazole/trimethoprim, norfloxacin, or ciprofloxacin for the prevention of recurrent SBP. Fluoroquinolones as a class have had increased black box warnings in recent years, making ciprofloxacin fall out of favor for long-term prophylaxis.5 Sulfamethoxazole/trimethoprim is extensively metabolized by the liver and is contraindicated in marked liver impairment.8 Therefore, it is necessary to search for a prophylaxis alternative with similar efficacy and a better safety profile.

Doxycycline is a broad-spectrum antibiotic that covers Gram-positive bacteria, including Streptococcus spp., resistant strains of Staphylococcus and Enterococcus, and Gram-negative bacteria, including Enterobacteriaceae. One randomized trial in cirrhotic patients with a previous episode of SBP showed that doxycycline was associated with a reduction in inflammatory markers, such as interleukin-6 and C-reactive protein, suggesting potential benefits of doxycycline in this patient population.7 At Methodist Dallas Medical Center (MDMC) and the Liver Institute at MDMC, doxycycline has been utilized for both primary and secondary prevention of SBP. In order to compare doxycycline with guideline-directed therapies for SBP prevention in cirrhotic patients, a retrospective, cohort study was designed to review patients who meet the criteria from July 2014 to July 2018. This study aims to compare the efficacy of doxycycline with that of guideline recommended therapies for primary and secondary SBP prophylaxis, the safety of doxycycline with that of guideline recommended therapies for primary and secondary SBP prophylaxis, and identify the association between chemoprophylaxis and the risk of infections from multidrug resistant organisms (MDROs) in SBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year-old with refractory ascites who are candidates for SBP prophylaxis per clinician's decision
* Patients diagnosed with cirrhosis based on clinical criteria
* Patients with a diagnosis of SBP confirmed by paracentesis

Exclusion Criteria:

* Patients who have secondary peritonitis other than SBP
* Patients who have a history of liver transplant prior to the initial episode of SBP
* Patients with incomplete medical records

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at MDMC at the Liver Institute Clinic with a diagnosis of SBP based on ascitic fluid PMN count greater than 250 cells/mm3 from July 2014 to July 2018.
Sampling Method: Non-Probability Sample
Enrollment: 841 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of reported SBP | July 2014 to July 2018
  Occurrence of reported SBP within 1-year of chemoprophylaxis initiation

SECONDARY OUTCOMES:
Incidences of death | July 2014 to July 2018
  Incidences of death within 1-year of chemoprophylaxis initiation
Incidences of Liver transplant | July 2014 to July 2018
  Incidences of liver transplant within 1-year of chemoprophylaxis initiation
Incidences of bacteremia | July 2014 to July 2018
  Incidences of bacteremia within 1-year of chemoprophylaxis initiation
Hospitalizations and ED visits due to AKI | July 2014 to July 2018
  Hospitalizations and ED visits due to AKI within 1-year of chemoprophylaxis initiation
Hospitalizations and ED visits due to Clostridioides difficile infection | July 2014 to July 2018
  Hospitalizations and ED visits due to Clostridioides difficile infection within 1-year of chemoprophylaxis initiation
Hospitalizations and ED visits due to diarrhea | July 2014 to July 2018
  Hospitalizations and ED visits due to diarrhea within 1-year of chemoprophylaxis initiation
Hospitalizations and ED visits due to hyperkalemia | July 2014 to July 2018
  Hospitalizations and ED visits due to hyperkalemia within 1-year of chemoprophylaxis initiation
Rate of infection with MDRO | July 2014 to July 2018
  Rate of infection with MDRO within 1-year of chemoprophylaxis initiation

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Rago, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided